CLINICAL TRIAL: NCT05701280
Title: Rehab With Electrical Stimulation Therapy to Optimize Rehabilitation Effect (RESTORE): A Pivotal Study
Brief Title: Pilot/Pivotal Study of DBS+Rehab After Stroke
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enspire DBS Therapy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDD 0084
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: Ischemic Stroke; Deep Brain Stimulation; DBS; Physical Therapy; Rehabilitation; Brain Stimulation
MeSH Terms: conditions — Stroke; Paresis; Ischemic Stroke | interventions — Deep Brain Stimulation; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, parallel study with partial crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Care Providers (Therapists), Investigators, and Outcome Assessors do not know to which group the participants are randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DBS+Rehab (Experimental): Active-DBS combined with motor rehabilitation
  Interventions: Device: Deep Brain Stimulation
- Rehab (Active Comparator): Control-DBS combined with motor rehabilitation
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation (DBS) of the dentate nucleus area of the cerebellum plus motor rehabilitation to improve upper-extremity function.
  Arms: DBS+Rehab
Other: Rehabilitation — Motor rehabilitation to improve upper-extremity function.
  Arms: Rehab

SUMMARY:
The RESTORE Stroke Study will evaluate the safety and effectiveness of DBS+Rehab for treating arm weakness and reduced function after a stroke.

DETAILED DESCRIPTION:
The RESTORE Stroke Study combines two phases of study under one protocol (pilot/pivotal). The first phase has a sample size of 40 subjects. The second phase has an estimated sample size of 162 subjects which may be adjusted based on analysis of the first phase.

Each subject will be implanted with the DBS system, undergo DBS program optimization, and be randomized to test treatment (Tt) or active-control treatment (Ct). After randomization, all subjects will participate in a five-month outpatient rehabilitation therapy program. After five months of blinded randomized testing, subjects assigned to active-control treatment (Ct) will cross over to receive test treatment (Tt) and participate in a second five-month therapy program.

ELIGIBILITY:
Key Inclusion Criteria:

* Ischemic stroke, with an initial incident occurring between 12 months to 6 years before implant, resulting in residual upper extremity hemiparesis.

Key Exclusion Criteria:

* Previous or subsequent cerebrovascular events resulting in residual upper extremity impairment
* Brain lesions with significant involvement of the brainstem, cerebellum, or thalamus

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment, Upper Extremity sub-scale (FMA-UE) | Week-12 to Week-32
  The change in FMA-UE is significantly greater for subjects who receive Test treatment (Tt) than Control treatment (Ct).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment, Upper Extremity sub-scale (FMA-UE) | Week-12 to Week-32
  The change in FMA-UE for subjects who receive Test treatment (Tt) is significantly above a clinically important difference (CID)

OTHER OUTCOMES:
Fugl-Meyer Assessment, Upper Extremity sub-scale (FMA-UE) | Week-32, Week-40 and Week 52
  Exploratory endpoints will be examined for the group originally assigned to Control treatment after crossover.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Barrow Neurological Institute (BNI), Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina